CLINICAL TRIAL: NCT00620685
Title: A 4-Week, Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Safety And Pharmacokinetic Profile Of 1 And 5 Mg Ph-797804 Administered Once Daily In Subjects With Rheumatoid Arthritis Who Are Taking Oral Methotrexate
Brief Title: A Study To Evaluate The Safety And Pharmacokinetic Profile Of A P38 Inhibitor (PH-797804) In Subjects With Rheumatoid Arthritis Who Are Also Taking Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A6631005
Record Dates: First submitted 2008-01-10; First posted 2008-02-21 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — PH 797804

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: PH-797804
- 3 (Experimental)
  Interventions: Drug: PH-797804

INTERVENTIONS:
Drug: Placebo — Tablet, once daily for 4 weeks
  Arms: 1
Drug: PH-797804 — Tablet, 1 mg PH-797804, once daily for 4 weeks
  Arms: 2
Drug: PH-797804 — Tablet, 5 mg PH-797804, once daily for 4 weeks
  Arms: 3

SUMMARY:
The hypothesis of this study is that the p38 inhibitor (PH-797804) will be safe and well tolerated in subjects with rheumatoid arthritis who are taking methotrexate and will not effect the blood levels of methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Adult with RA for at least 6 months
* Stable weekly dosage of oral methotrexate 12.5- 25 mg/week

Exclusion Criteria:

* Severe, progressive and/or uncontrolled other disease
* Chronic or recent serious infection; current infection
* Concomitant use of RA therapy other than methotrexate with some exceptions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory data, vital signs, 12-lead ECGs and physical examination findings | 6 weeks

SECONDARY OUTCOMES:
Estimate the effects of multiple doses of PH-797804 on the pharmacokinetic profile of methotrexate in subjects with RA taking a stable dose of MTX | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Bingham Farms, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Duncansville, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631005